CLINICAL TRIAL: NCT01524965
Title: The Effect of the Timing of Postoperative Mobilisation After Locking Plate Osteosynthesis of Fractures of the Surgical Neck of the Humerus.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment decline due to change in clinical practice to less surgery for the fractures of interest
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government)
Responsible Party: Principal Investigator, Tuomas Lahdeoja, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS-272/13/03/02/2010
Record Dates: First submitted 2012-01-22; First posted 2012-02-02 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Humeral Fracture
Keywords: Locking Plate; Physiotherapy
MeSH Terms: conditions — Humeral Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate mobilisation (Experimental)
  Interventions: Procedure: Immediate mobilisation after locking-plate osteosynthesis; Device: Osteosynthesis with a locking plate (Philos)
- Standard mobilisation (Active Comparator)
  Interventions: Procedure: Standard mobilisation after locking plate osteosynthesis; Device: Osteosynthesis with a locking plate (Philos)

INTERVENTIONS:
Procedure: Immediate mobilisation after locking-plate osteosynthesis — Immediate passive range of motion exercises are begun postoperatively, after 3 weeks, active unloaded mobilisation begins after three weeks and active, loaded use is allowed 6 weeks postoperatively.
  Surgical procedure is open reduction of the fracture and internal fixation of the fracture using a locking plate using standard deltopectoral approach and AO principles in fracture management.
  Arms: Immediate mobilisation
Procedure: Standard mobilisation after locking plate osteosynthesis — Immediately postoperatively the arm is held in a sling, active mobilisation of healthy joints and pendel exercises are befun. Passive range of motion exercises of the shoulder are begun 3 weeks postoperatively. Active mobilisation begins after six weeks.
  Surgical procedure is open reduction of the fracture and internal fixation of the fracture using a locking plate using standard deltopectoral approach and AO principles in fracture management.
  Arms: Standard mobilisation
Device: Osteosynthesis with a locking plate (Philos) — Standard open reduction and internal fixation using a deltopectoral approach. Fracture fixation is done using a locking plate (Philos, Synthes) following the AO principles of fracture management.

SUMMARY:
Open reduction and locking plate osteosynthesis is a commonly used and well-accepted treatment for displaced fractures of the proximal humerus. The shoulders tend to end stiff despite intensive rehabilitation, limiting the function of the upper extremity and decreasing the quality of life. The accepted postoperative mobilisation protocol includes passive exercises until six weeks postoperatively and active range of motion exercises after that. There is good evidence that conservatively treated fractures of the same site heal better and faster if mobilised immediately. The study compares "standard mobilisation" versus "immmediate mobilisation" in a prospective, randomized, controlled trial in order to find the optimal time-frame for physiotherapy to produce best possible results. Outcome measures are assessed at specific time points after the operation and comparisons between groups are made to follow the rate of recovery and end results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Surgery can be performed within 10 days of injury
* A dislocated (>1cm or 35 degrees) AO 11-A2, -A3, -B1 or -B2 fracture of the surgical neck of the proximal humerus with a possible fracture of the Tuberculum Majus

Exclusion Criteria:

* Glenohumeral dislocation
* Fracture of the Tuberculum Minus
* Open fracture
* Additional fractures in the shoulder region
* Other injuries requiring surgical treatment
* Clinically significant injury of the brachial plexus or vasculature
* Pathological fracture associated with cancer
* History of a fracture of the clavicle, scapula or humerus, or history of a very significant disease or trauma of the shoulder region (hemiparesis, tumour, osteomyelitis, grave arthrosis etc)
* Rheumatoid Arthritis in the shoulder requiring active treatment
* Reduced co-operation or incapability for independent living (dementia, mental illness, drug- or alcohol abuse etc)
* Unwillingness to accept some of the treatment options.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-05; Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Disablities of Arm, Hand and Shoulder | 3 weeks
  Validated patient-reported upper extremity function scale
Disablities of Arm, Hand and Shoulder | 6 weeks
  Validated patient-reported upper extremity function scale
Disablities of Arm, Hand and Shoulder | 3 months
  Validated patient-reported upper extremity function scale
Disablities of Arm, Hand and Shoulder | 6 months
  Validated patient-reported upper extremity function scale
Disablities of Arm, Hand and Shoulder | 1 year
  Validated patient-reported upper extremity function scale
Disablities of Arm, Hand and Shoulder | 2 years
  Validated patient-reported upper extremity function scale

SECONDARY OUTCOMES:
Constant Score | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  subjective and objective shoulder score
Simple Shoulder Test (SST) | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  another shoulder score
Pain in rest and motion (2 different values) | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Numeric rating scale 0-10
Subjective satisfaction | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Patient reported, Numeric Rating Scale 0-10
Quality of Life | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Using the 15D instrument
Complications | 3 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years
  Complications of surgery and postoperative phase

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Lähdeoja, MD, Principal Investigator — Helsinki University Central Hospital; Mika Paavola, MD, PhD, Study Director — Helsinki University Central Hospital; Jarkko Pajarinen, MD, PhD, Study Director — Helsinki University Central Hospital; Seppo Koskinen, Study Chair — Helsinki University Central Hospital; Antti Malmivaara, MD, PhD, Study Chair — Finnish Institute for Health and Welfare; Reijo Sund, MD, PhD, Study Chair — Finnish Institute for Health and Welfare
Locations (1):
- Töölö Hospital, Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196